CLINICAL TRIAL: NCT04257279
Title: Prospective Robotic Global Research Study (PROGRESS)
Acronym: PROGRESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Globus Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGC18-002
Record Dates: First submitted 2019-04-29; First posted 2020-02-06 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Lumbar Disc Disease
Keywords: spine
MeSH Terms: conditions — Intervertebral disc disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Robotic (Experimental): Patients receiving spine surgery with posterior stabilization placed by ExcelsiusGPS
  Interventions: Procedure: ExcelsiusGPS™

INTERVENTIONS:
Procedure: ExcelsiusGPS™ — The ExcelsiusGPS™ is a Robotic Positioning System that includes a computer controlled robotic arm, hardware, and software that enables real time surgical navigation and robotic guidance using radiological patient images (pre-operative CT, intra-operative CT and fluoroscopy), using a dynamic reference base and positioning camera.

SUMMARY:
The purpose of this study is to prospectively review outcomes of patients who have surgery with the ExcelsiusGPS™ robotics system in order to analyze screw placement accuracy. Patient demographics, intraoperative data and radiographic imaging to determine screw placement accuracy will be collected and reviewed. This information will be compared in a separate study to retrospectively collected data from sites who have done a similar number of cases without the robot.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and a maximum age of 85 years
* Require surgery that includes posterior stabilization with screws to be inserted in cervical, thoracic, lumbar spine or sacrum
* Able to sign Informed Consent

Exclusion Criteria:

* Previous fusion or fusion attempt at index level(s)
* DEXA score of -2.5 or below (only if clinically indicated - optional)
* Presence of a disease entity or condition which totally precludes possibility of bony fusion (e.g. metastatic cancer, HIV, long term use of steroids, etc.)
* History of substance abuse (drugs or alcohol)
* Mentally incompetent or prisoner
* Worker's compensation
* Pregnant or intention to become pregnant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale | Baseline
  Pain rating scale
Numeric Rating Scale | 2 weeks
  Pain rating scale
Numeric Rating Scale | 3 months
  Pain rating scale
Numeric Rating Scale | 6 months
  Pain rating scale
Numeric Rating Scale | 12 months
  Pain rating scale
Numeric Rating Scale | 24 months
  Pain rating scale
Oswestry Disability Index | Baseline
  Index derived from the Oswestry Low Back Pain Questionnaire
Oswestry Disability Index | 2 weeks
  Index derived from the Oswestry Low Back Pain Questionnaire
Oswestry Disability Index | 3 months
  Index derived from the Oswestry Low Back Pain Questionnaire
Oswestry Disability Index | 6 months
  Index derived from the Oswestry Low Back Pain Questionnaire
Oswestry Disability Index | 12 months
  Index derived from the Oswestry Low Back Pain Questionnaire
Oswestry Disability Index | 24 months
  Index derived from the Oswestry Low Back Pain Questionnaire
SF-12 | Baseline
  12-Item short form health survey
SF-12 | 2 weeks
  12-Item short form health survey
SF-12 | 3 months
  12-Item short form health survey
SF-12 | 6 months
  12-Item short form health survey
SF-12 | 12 months
  12-Item short form health survey
SF-12 | 24 months
  12-Item short form health survey
Screw Placement Accuracy | 2 weeks
  Gertzbein Robbins Scale for screw accuracy
Complications | through study completion, 2 years
  Adverse Event

CONTACTS AND LOCATIONS:
Locations (1):
- Southeastern Spine Institute, Mt. Pleasant, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No